CLINICAL TRIAL: NCT06169397
Title: A Long-term Multicenter Open-label Study to Evaluate the Long-term Safety and Durability of Effect of XTMAB-16 in Patients With Pulmonary Sarcoidosis With or Without Extra-pulmonary Involvement
Brief Title: An Open-label Extension Study of XTMAB-16 in Patients With Pulmonary Sarcoidosis
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Xentria, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XTMAB-16-202
Record Dates: First submitted 2023-11-17; First posted 2023-12-13 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Sarcoidosis
MeSH Terms: conditions — Sarcoidosis, Pulmonary

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- XTMAB-16 Treatment (Experimental): Dose to be established in the XTMAB-16-201 Study.
  Interventions: Drug: XTMAB-16

INTERVENTIONS:
Drug: XTMAB-16 — XTMAB-16 infusion

SUMMARY:
Open-label Study to Evaluate the Long-term Safety and Durability of Effect of XTMAB-16 in Patients With Pulmonary Sarcoidosis With or Without Extra-pulmonary Involvement

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study if the following criteria apply:

* Completion of XTMAB-16-201 study: completion of Week 12 (Part A) or Week 24 (Part B) assessments.
* Participants from XTMAB-16-201 Part A and Part B should be on a stable steroid dose for at least 2 weeks prior to informed consent/Day 1 of XTMAB-16-202 (Day 1 should occur at the next scheduled dosing visit on the assigned dose frequency cohort of XTMAB 16 201 ± 2 weeks).

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Evidence of treatment-related AEs requiring treatment discontinuation per XTMAB-16-201 protocol observed in XTMAB-16-201 study.
* Evidence of treatment failure observed in XTMAB-16-201 study per protocol definition.
* Pregnant or breastfeeding women or women who are planning to be pregnant during the course of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Adverse Events (AEs), including Serious Adverse Events (SAEs), and Adverse Events of Special Interests (AESIs) throughout the study duration | Through study completion, an average of 4 years

SECONDARY OUTCOMES:
Durability/maintenance of effect of XTMAB-16 as characterized by corticosteroid dosing (maintain or lower steroid dosing) | Through study completion, an average of 4 years
Durability/maintenance of effect of XTMAB-16 as characterized by changes in quality of life measured by Kings Sarcoidosis Questionnaire Lung | Through study completion, an average of 4 years
Durability/maintenance of effect of XTMAB-16 as characterized by changes in quality of life measured by Kings Sarcoidosis Questionnaire General | Through study completion, an average of 4 years
Durability/maintenance of effect of XTMAB-16 as characterized by changes in quality of life measured by Leicester Cough Questionnaire | Through study completion, an average of 4 years
Durability/maintenance of effect of XTMAB-16 as characterized by changes in quality of life measured by Steroid Toxicity Questionnaire | Through study completion, an average of 4 years
Durability/maintenance of effect of XTMAB-16 measured by Pulmonary Function Test (forced vital capacity) | Through study completion, an average of 4 years
Immunogenicity (number of participants who test positive for anti drug antibodies and/or neutralizing antibodies) in the context of long-term dosing | Through study completion, an average of 4 years
Long-term effect of XTAMB-16 on serum biomarkers important to cytokine pathway and granuloma formation (ACE, IL-6, sIL-2R, sTNFa, CRP, IL-1b, calcitriol) in sarcoidosis | Through study completion, an average of 4 years

CONTACTS AND LOCATIONS:
Locations (11):
- United States (5):
  - Xentria Investigative Site, Denver, Colorado
  - Xentria Investigative Site, Chicago, Illinois
  - Xentria Investigative Site, Greenville, North Carolina
  - Xentria Investigative Site, Cincinnati, Ohio
  - Xentria Investigative Site, Philadelphia, Pennsylvania
- Xentria Investigative Site, Prague, Czechia
- Xentria Investigative Site, Bielsk Podlaski, Poland
- United Kingdom (4):
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry, England
  - King's College Hospital NHS Foundation Trust, London, England
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, England
  - NHS Tayside, Perth, Scotland